CLINICAL TRIAL: NCT01618240
Title: Determining Predictors of Adequate Upper Airway Function in Long-term Ventilated Patients
Brief Title: Predictors of the Ability to Protect the Airway in Long-term Ventilated Patients
Status: Completed | Type: Observational
Sponsor: Massachusetts General Hospital (Other)
Responsible Party: Principal Investigator, Matthias Eikermann, Assistant Professor, Massachusetts General Hospital
Other Study IDs: 2010P001919A
Record Dates: First submitted 2012-06-06; First posted 2012-06-13 (Estimated); Results first posted 2013-08-27 (Estimated); Last update posted 2014-10-13 (Estimated); Status verified 2013-05

CONDITIONS: Swallowing Disorder; Aspiration; Long Term Ventilation
Keywords: FEES; PAS; VPSR; MRC
MeSH Terms: conditions — Deglutition Disorders | interventions — Ventilators, Mechanical

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Whole Blood
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (1):
- Long term ventilated subjects: Muscle Strength Measurement, ventilator
  Interventions: Other: Muscle Strength Measurement; Other: Ventilator

INTERVENTIONS:
Other: Muscle Strength Measurement — MRC score (0-60) is a clinical assessment of muscle power on abduction of the arm, flexion of the forearm, extension of the wrist, flexion of the leg, extension of the knee and dorsal flexion of the foot with the score of (0-5) on each measurement
Other: Ventilator — A mechanical ventilator is used to assist or replace spontaneous breathing.

SUMMARY:
First part of a 2 part study with the same IRB protocol #, and labeled 'A'. Investigators hypothesized that clinical muscle strength assessment (manual muscle testing) predicts the ability to protect the airway during swallowing in long-term ventilated subjects. More specifically, the investigators hypothesized that low muscle strength is associated with the inability to clear secretions from the peri-laryngeal area (valleculae and pyriform sinus residue scale (VPSR scale [NRS: 0-4] of > 1) and entering the materials into airway (PAS scale [1-8]> 1), which should predispose to endotracheal aspiration.

ELIGIBILITY:
Inclusion Criteria:

1. Patients admitted to the Respiratory Acute Care Unit and Surgical Intensive Care Unit, units with a mixed collection of long term ventilated patients in a major academic teaching hospital.
2. Age over 18 years.
3. Long-term ventilated patients (>10 days) with tracheotomies

Exclusion Criteria:

1. Decreased level of consciousness as defined by a Richmond Agitation Sedation Scale (RASS) of 0.
2. Non-cooperative patient, CAM score positive for delirium.
3. For women: pregnancy.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Long term ventilated and tracheostomized patients in the Respiratory Acute and Surgical Intensive Care Unit
Sampling Method: Non-Probability Sample
Enrollment: 30 (Actual)
Dates: Start 2011-01; Primary Completion 2012-04 (Actual); Study Completion 2012-04 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Matthias Eikermann, MD, PhD, Principal Investigator — MGH, Harvard Medical School
Locations (1):
- Massachusetts general Hospital, Boston, Massachusetts, United States

REFERENCES:
- [Background] Rosenbek JC, Robbins JA, Roecker EB, Coyle JL, Wood JL. A penetration-aspiration scale. Dysphagia. 1996 Spring;11(2):93-8. doi: 10.1007/BF00417897. PMID 8721066
- [Background] Butler SG, Stuart A, Markley L, Rees C. Penetration and aspiration in healthy older adults as assessed during endoscopic evaluation of swallowing. Ann Otol Rhinol Laryngol. 2009 Mar;118(3):190-8. doi: 10.1177/000348940911800306. PMID 19374150
- [Background] Kleyweg RP, van der Meche FG, Schmitz PI. Interobserver agreement in the assessment of muscle strength and functional abilities in Guillain-Barre syndrome. Muscle Nerve. 1991 Nov;14(11):1103-9. doi: 10.1002/mus.880141111. PMID 1745285
- [Result] Mirzakhani H, Williams JN, Mello J, Joseph S, Meyer MJ, Waak K, Schmidt U, Kelly E, Eikermann M. Muscle weakness predicts pharyngeal dysfunction and symptomatic aspiration in long-term ventilated patients. Anesthesiology. 2013 Aug;119(2):389-97. doi: 10.1097/ALN.0b013e31829373fe. PMID 23584384

RESULTS

PARTICIPANT FLOW:
Groups:
- Long-term Ventilated Subjects: Long-term (>10 days hours) ventilated subjects were included.
Period: Overall Study
Arm/Group | Long-term Ventilated Subjects
Started | 30
Completed | 30
Not Completed | 0

BASELINE CHARACTERISTICS:
Population: 30 long-term ventilated subjects were included (ventilated > 10 days). Subjects had a Richmond Agitation Sedation score of >0, had no delirium, had no abnormalities of the larynx or pharynx, and no history of chemotherapy or radiotherapy to the head/ neck, or of degenerative neurological disease.
Groups:
- Baseline Population: Thirty long-term ventilated patients admitted in two intensive care units at Massachusetts General Hospital.
Arm/Group | Baseline Population
Number analyzed (Participants) | 30
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 23
  >=65 years | 7
Age, Continuous [Mean (Standard Deviation); unit: years] | 55 (14)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 14
  Male | 16
Region of Enrollment [Number; unit: participants]
  United States | 30

OUTCOME MEASURES:

1. Primary Outcome: Muscle Strength
Description: We use Medical Research Council (MRC) scale (0-60) to evaluate the degree of muscle weakness in the tracheostomized patients.
Time Frame: Within 24 hours of fiberoptic endoscopic evaluation of swallow
Measure: Number; unit: participants
Groups:
- Muscle Strength Measurement: Muscle Strength Measurement : MRC score (0-60) is a clinical assessment of muscle power on abduction of the arm, flexion of the forearm, extension of the wrist, flexion of the leg, extension of the knee and dorsal flexion of the foot with the score of (0-5) on each measurement
Arm/Group | Muscle Strength Measurement
Number analyzed (Participants) | 30
participants
  Clinically significant muscle weakness (<48) | 20
  No clinically significant muscle weakness (>=48) | 10

2. Secondary Outcome: Number of Patients With Muscle Weakness (MRC<48) Who Developed Clinical Aspiration
Time Frame: Within 3 month follow-up
Measure: Number; unit: participants
Arm/Group | Muscle Strength Measurement
Number analyzed (Participants) | 20
participants
  Symptomatic aspiration | 14
  No symptomatic aspiration | 6

ADVERSE EVENTS:
Groups:
- Long-term Ventilated Subjects: 30 consented long-term ventilated patients
Arm/Group | Long-term Ventilated Subjects
Serious Adverse Events (participants affected / at risk) | 0/30
Other Adverse Events (participants affected / at risk) | 0/30

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes